CLINICAL TRIAL: NCT00169299
Title: Herbal Alternatives for Menopause Symptoms: A Randomized Trial
Brief Title: Herbal Alternatives for Menopause Symptoms (HALT Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AG017057 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Vasomotor Symptoms Associated With Menopause
Keywords: Menopause; Vasomotor; Black cohosh; Herbs; Hot flashes; HT; CAM
MeSH Terms: conditions — Hot Flashes | interventions — black cohosh root extract

INTERVENTIONS:
Drug: Black cohosh
Drug: Multibotanical preparation
Drug: Multibotanical preparation + dietary soy counseling
Drug: Conjugated equine estrogen +/- medroxyprogesterone acetate

SUMMARY:
Surveys indicate that 25 to 33% of women have moderate to severe menopausal symptoms including hot flashes, night sweats, and disturbed sleep. The treatment of choice in the medical community for these symptoms is hormone replacement therapy, which is estrogen and sometimes progestin. Many women also use over-the-counter herbal remedies. However, less is known about how well these products work, or their safety. Few have undergone the kind of rigorous testing required of prescription drugs and little is known about their long-term effectiveness in relieving symptoms.

The purpose of this study is to compare several over-the-counter herbal remedies to hormone replacement therapy. Our primary aim is to look at the effects of these remedies on your self-reported menopausal symptoms. We will also be measuring their effects on other factors known to be affected by hormone replacement therapy: cholesterol, blood sugar, bone density, vaginal cell structure, and blood clotting.

DETAILED DESCRIPTION:
Hormone replacement therapy (HT: estrogen and progestin) remains the treatment of choice for women with vasomotor symptoms, and long-term HT has been recommended for prevention purposes. The demand for alternatives to HT, and the availability and use of over-the-counter products including dietary phytoestrogen supplements, and naturopathic medicines has grown dramatically. Few of these products have faced the rigors of randomized trials and none have been tested to evaluate their effects on long-term outcomes.

The purpose of this 4-year, randomized controlled trial is to evaluate the efficacy and safety of three alternative approaches utilizing phytoestrogens to treat vasomotor symptoms in peri- and postmenopausal women. The treatments were chosen because of the scientific evidence supporting a possible benefit, the availability of products with adequate quality control, their frequency of use in naturopathic medicine, and our ability to blind participants to the intervention. The 5 proposed treatment arms are: 1) conjugated equine estrogen with or without medroxyprogesterone acetate in women with or without an intact uterus respectively; 2) a single herbal product, black cohosh; 3) a multibotanical preparation; 4) a combination regimen that includes the same multibotanical preparation plus soy diet counseling; and 5) placebo. Our primary aim is to compare the effects of three alternative treatments, HRT and placebo on the frequency and intensity of vasomotor symptoms measured by The Wiklund Menopause Symptom Checklist and a daily Vasomotor Symptom Diary. Our secondary aims are to compare the effects of three alternative treatments, HRT and placebo on: 1) vaginal cytology (vaginal maturation index); 2) serum lipids (total cholesterol, HDL and LDL cholesterol, triglycerides); 3) bone mineral density (hip and spine dual energy x-ray absorptiometry scan); 4) glucose metabolism (insulin, fasting blood glucose); and 5) coagulation factors (fibrinogen, PAI-1).

Our hypotheses are that compared to placebo, the three alternative treatments tested in this proposal will; reduce frequency of hot flashes and night sweats, improve vaginal maturation and decrease vagina atrophy as measured by maturation index, lower total cholesterol and LDL with no effect on HDL, reduce the rate of decline in bone mineral density (BMD), and have no effect on glucose metabolism or clotting factors.

To accomplish our specific aims we will: 1) recruit and randomize approximately peri- and post-women to one of 5 treatment arms for one year; 2) collect measurements of primary and secondary outcomes at baseline, 3, 6, and 12 months; and 3) compare changes in outcomes in the groups taking alternative treatments to those in the HRT and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 45 - 55
* peri- or post-menopausal
* moderate to severe vasomotor symptoms
* normal thyroid stimulating hormone
* proof of normal mammogram within past 2 years

Exclusion Criteria:

* use of HT or oral contraceptives within past 3 months
* use of herbs or alternative or complementary medicines for vasomotor symptoms within past 1 month
* medical history of contraindications to HT
* bone mineral density greater than 2 standard deviations below age specific mean
* bilateral oophorectomy
* current use of tamoxifen, raloxifene, bisphosphonates, cholesterol-lowering medications, prescription blood-thinners, or oral steroids
* pregnant or planning to become pregnant
* allergy to soybeans or soy protein
* unable to swallow pills
* current participation in another investigational drug trial
* intention to move out of area in the next 12 months
* non-compliance with procedures involved in screening and run-in trial

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 351
Dates: Start 2001-06; Study Completion 2004-09

PRIMARY OUTCOMES:
Self report daily diary of frequency and intensity of vasomotor symptoms at BL, 3, 6 and 12 months.
Wiklund Menopause Symptom Checklist at BL, 3, 6 and 12 months.

SECONDARY OUTCOMES:
Vaginal cytology (vaginal maturation index)at BL, 3 and 12 months.
Serum lipids (total cholesterol, HDL and LDL cholesterol, triglycerides) at BL, 3, 6, and 12 months.
Bone mineral density (hip and spine dual energy x-ray absorptiometry scan) at BL, 6 and 12 months.
Glucose metabolism (insulin, fasting blood glucose) at BL, 3, 6, and 12 months.
Coagulation factors (fibrinogen, PAI-1) at BL, 3, 6, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Newton, PhD, Principal Investigator — Group Health Cooperative, Center for Health Studies
Locations (1):
- Group Health Cooperative, Center for Health Studies, Seattle, Washington, United States

REFERENCES:
- [Derived] Newton KM, Reed SD, LaCroix AZ, Grothaus LC, Ehrlich K, Guiltinan J. Treatment of vasomotor symptoms of menopause with black cohosh, multibotanicals, soy, hormone therapy, or placebo: a randomized trial. Ann Intern Med. 2006 Dec 19;145(12):869-79. doi: 10.7326/0003-4819-145-12-200612190-00003. PMID 17179056